CLINICAL TRIAL: NCT02430051
Title: Sensory Adapted Dental Environments to Enhance Oral Care for Children (SADE-2)
Brief Title: Sensory Adapted Dental Environments to Enhance Oral Care for Children
Acronym: SADE-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Sharon Cermak, Professor, University of Southern California
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DE024978-01
Record Dates: First submitted 2015-04-24; First posted 2015-04-29 (Estimated); Results first posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Autism
Keywords: sensory processing; oral care; electrodermal activity; cooperation; anxiety; distress; stress; behavior; occupational therapy
MeSH Terms: conditions — Autistic Disorder; Anxiety Disorders; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Regular Dental Environment (No Intervention): There are two dental environments - the regular dental environment and the sensory dental environment; each child will be randomized to which is first. In the Regular dental environment no sensory characteristics of the dental environment are altered, the cleaning is conducted as per usual.
- Sensory Adapted Dental Environment (Experimental): In the Sensory Adapted Dental Environment the sensory characteristics of the dental environment are altered (visual, auditory, and tactile adaptations).
  Interventions: Behavioral: Sensory Adapted Dental Environment

INTERVENTIONS:
Behavioral: Sensory Adapted Dental Environment — The SADE intervention includes adaptations such as dimmed lighting, moving projections on the ceiling (fish, bubbles), exposure to soothing music, and application of a butterfly vest with wings that wrap around the child to provide calming sensations.
  Other Names: SADE Intervention
  Arms: Sensory Adapted Dental Environment

SUMMARY:
The goal of this project is to examine the efficacy of a sensory adapted dental environment (SADE) for children who have difficulty tolerating oral care in the dental clinic. The investigators hypothesize that adapting the sensory environment in the dental office by modifying the sounds, sights,and tactile experiences will result in decreased anxiety, increased cooperation, and fewer behavior problems for children with Autism Spectrum Disorders (ASD). This has the potential to contribute to increased child comfort as well as safer, more efficient, and less costly treatment for a large population, as potentially more than one-fourth of all children may benefit from a sensory adapted dental environment.

DETAILED DESCRIPTION:
This project, which builds upon the investigator's previous R34 National Institute of Dental and Craniofacial Research (NIDCR) Planning and Feasibility study, is designed to examine the efficacy of a sensory adapted dental environment (SADE) to enhance oral care for children with autism spectrum disorders (ASD). Children with ASD often exhibit sensory over-responsivity when confronted with experiential aspects of dental visits such as exposure to bright fluorescent lighting, touch in or around the mouth, or the texture and smell of various oral care products. This often results in increased anxiety and negative behavioral responses which hinder the dentist's ability to perform treatment. In the proposed project, the investigators test a SADE intervention designed to reduce children's anxiety and negative responses during oral care.

The SADE intervention includes adaptations such as dimmed lighting, moving projections on the ceiling (fish, bubbles), exposure to soothing music, and application of a butterfly vest with wings that wrap around the child to provide calming sensations.

The specific aims are to conduct a randomized clinical trial in order to:

1. Determine if SADE, relative to a regular dental environment (RDE), reduces physiological anxiety and negative responses (behavioral distress, perception of pain, sensory discomfort) during dental cleaning for children with ASD.
2. Identify whether physiological anxiety mediates the beneficial effects of the intervention and whether severity of ASD and communication ability, or dental anxiety, sensory over-responsivity, and age act as moderating variables.
3. Assess the quality of care and cost effectiveness/savings of the dental cleaning associated with SADE.

Research participants will be 220 ethnically diverse children aged 6-12 years. Using a randomized counterbalanced study design, each child will undergo two dental cleanings four months apart: one dental cleaning in RDE and one dental cleaning in SADE.

This project is significant because it is the first full-scale trial of an intervention designed to reduce oral care problems in children with ASD. It is theoretically important because it will elucidate the mechanisms that underlie the effects of the SADE intervention. Based on the study findings, the investigators will develop a model to transform the standard of pediatric dental care by modifying the sensory qualities of the dental environment. This model will have the potential to be utilized in dental clinics worldwide. As such, the project promises to have a major public health impact insofar as the potential gains in oral health, child comfort, and cost-savings will be dramatic, potentially applying to more than one-fourth of all children.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of autism using ADOS;
* Parents speak English or Spanish;
* Have experienced at least one prior dental cleaning;
* In need of an oral cleaning (no previous cleaning within past four months).

Exclusion Criteria:

* Cleft palate or other oral condition which makes dental care more difficult than usual practice;
* Prescription of anti-cholinergic drugs (which may alter EDA);
* Presence of orthodontia (braces);
* Significant motor impairment, such as cerebral palsy;
* Any known genetic, endocrine, or metabolic dysfunctions;
* Participation in the R34 SADE pilot study;
* Any medical condition such as significant cardiac problems that would place the individual at increased risk in the study.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 220 (Actual)
Dates: Start 2015-05; Primary Completion 2021-04-29 (Actual); Study Completion 2021-04-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Cermak, EdD, Principal Investigator — University of Southern California
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States

REFERENCES:
- [Background] Cermak SA, Stein Duker LI, Williams ME, Lane CJ, Dawson ME, Borreson AE, Polido JC. Feasibility of a sensory-adapted dental environment for children with autism. Am J Occup Ther. 2015 May-Jun;69(3):6903220020p1-10. doi: 10.5014/ajot.2015.013714. PMID 25871593
- [Background] Stein LI, Lane CJ, Williams ME, Dawson ME, Polido JC, Cermak SA. Physiological and behavioral stress and anxiety in children with autism spectrum disorders during routine oral care. Biomed Res Int. 2014;2014:694876. doi: 10.1155/2014/694876. Epub 2014 Jul 10. PMID 25114916
- [Background] Stein LI, Polido JC, Cermak SA. Oral care and sensory over-responsivity in children with autism spectrum disorders. Pediatr Dent. 2013 May-Jun;35(3):230-5. PMID 23756306
- [Background] Stein LI, Polido JC, Cermak SA. Oral care and sensory concerns in autism. Am J Occup Ther. 2012 Sep-Oct;66(5):e73-6. doi: 10.5014/ajot.2012.004085. PMID 22917131
- [Background] Stein LI, Polido JC, Najera SO, Cermak SA. Oral care experiences and challenges in children with autism spectrum disorders. Pediatr Dent. 2012 Sep-Oct;34(5):387-91. PMID 23211914
- [Background] Stein LI, Polido JC, Mailloux Z, Coleman GG, Cermak SA. Oral care and sensory sensitivities in children with autism spectrum disorders. Spec Care Dentist. 2011 May-Jun;31(3):102-10. doi: 10.1111/j.1754-4505.2011.00187.x. PMID 21592164
- [Derived] Stein Duker LI, Como DH, Jolette C, Vigen C, Gong CL, Williams ME, Polido JC, Florindez-Cox LI, Cermak SA. Sensory Adaptations to Improve Physiological and Behavioral Distress During Dental Visits in Autistic Children: A Randomized Crossover Trial. JAMA Netw Open. 2023 Jun 1;6(6):e2316346. doi: 10.1001/jamanetworkopen.2023.16346. PMID 37266941

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from health clinics (eg, CHLA dental clinic), community service providers (eg, developmental disability service providers, resource fairs), therapy and behavioral clinics, patient referrals, parent support groups, social media, and the Los Angeles Unified School District.
Groups:
- Regular Dental Environment First, Then Sensory Adapted Dental Environment: Dental Visit #1 (Day 5-95):
  Participants received their first dental cleaning in the Regular Dental Environment (RDE). In this condition, no sensory characteristics of the dental environment are altered and the cleaning is conducted in a standard manner (oral examination, prophylaxis, fluoride).
  Dental Visit #2 (Day 125-215):
  Participants received their second dental cleaning in the Sensory Adapted Dental Environment (SADE) approximately 6 months after their first dental cleaning. In the SADE, the sensory characteristics of the dental environment are altered (visual, auditory, tactile adaptations) including dimming lighting, moving projections on the ceiling, exposure to soothing music, and application of a butterfly vest with wings that wrap around the child to provide a calming sensation.
- Sensory Adapted Dental Environment First, Then Regular Dental Environment: Dental Visit #1 (Day 5-95):
  Participants received their first dental cleaning in the Sensory Adapted Dental Environment (SADE). In the SADE, the sensory characteristics of the dental environment are altered (visual, auditory, tactile adaptations) including dimming lighting, moving projections on the ceiling, exposure to soothing music, and application of a butterfly vest with wings that wrap around the child to provide a calming sensation.
  Dental Visit #2 (Day 125-215):
  Participants received their second dental cleaning in the Regular Dental Environment (RDE) approximately 6 months after their first dental cleaning. In this condition, no sensory characteristics of the dental environment are altered and the cleaning is conducted in a standard manner (oral examination, prophylaxis, fluoride).
Period: Overall Study
Arm/Group | Regular Dental Environment First, Then Sensory Adapted Dental Environment | Sensory Adapted Dental Environment First, Then Regular Dental Environment
Started | 83 | 80
Second Dental Visit | 70 | 68
Completed | 70 | 68
Not Completed | 13 | 12
Not completed — Withdrawal by Subject | 6 | 3
Not completed — Dropped due to not meeting scheduling requirements | 6 | 9
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Regular Dental Environment First, Then Sensory Adapted Dental Environment: Dental Visit #1 (Day 5-95) Participants received their first dental cleaning in the Regular Dental Environment (RDE). In this condition, no sensory characteristics of the dental environment are altered and the cleaning is conducted in a standard manner (oral examination, prophylaxis, fluoride).
  Dental Visit #2 (Day 125-215) Participants received their second dental cleaning in the Sensory Adapted Dental Environment (SADE) approximately 6 months after their first dental cleaning. In the SADE, the sensory characteristics of the dental environment are altered (visual, auditory, tactile adaptations) including dimming lighting, moving projections on the ceiling, exposure to soothing music, and application of a butterfly vest with wings that wrap around the child to provide a calming sensation.
- Sensory Adapted Dental Environment First, Then Regular Dental Environment: Dental Visit #1 (Day 5-95) Participants received their first dental cleaning in the Sensory Adapted Dental Environment (SADE). In the SADE, the sensory characteristics of the dental environment are altered (visual, auditory, tactile adaptations) including dimming lighting, moving projections on the ceiling, exposure to soothing music, and application of a butterfly vest with wings that wrap around the child to provide a calming sensation.
  Dental Visit #2 (Day 125-215) Participants received their second dental cleaning in the Regular Dental Environment (RDE) approximately 6 months after their first dental cleaning. In this condition, no sensory characteristics of the dental environment are altered and the cleaning is conducted in a standard manner (oral examination, prophylaxis, fluoride).
- Total: Total of all reporting groups
Arm/Group | Regular Dental Environment First, Then Sensory Adapted Dental Environment | Sensory Adapted Dental Environment First, Then Regular Dental Environment | Total
Number analyzed (Participants) | 70 | 68 | 138
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.19 (2.04) | 9.33 (1.93) | 9.26 (1.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 58 | 56 | 114
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 50 | 47 | 97
  Not Hispanic or Latino | 20 | 21 | 41
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 8 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 7 | 4 | 11
  White | 53 | 52 | 105
  More than one race | 6 | 3 | 9
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 70 | 68 | 138
Autism Diagnostic Observation Schedule-2 (ADOS-2) Severity Score [Mean (Standard Deviation); unit: score on a scale] — The ADOS-2 is a semi-structured, standardized performance-based observational assessment of social affect, communication, reciprocal social interaction, restricted and repetitive behaviors, imagination/creativity, stereotyped behaviors, and restricted interests. The severity (comparison) score is used as a standardized measure of autism symptom severity, independent of age and language level. The score ranges from 1 to 10, with higher scores indicating greater severity of autism-related symptoms (i.e., 3-4: low, 5-7: moderate, 8-10: high).
  score on a scale | 6.19 (1.78) | 6.65 (1.89) | 6.41 (1.84)
Wechsler Abbreviated Scale of Intelligence (WASI-II) Full Scale Intelligence Quotient (FSIQ4) [Mean (Standard Deviation); unit: score on a scale] — The WASI-II is a reliable and valid standardized measure of cognitive ability. The FSIQ-4 is derived from four subtests (Vocabulary, Similarities, Block Design, and Matrix Reasoning). The FSIQ-4 is calculated by summing the scaled scores from all four subtests and converting the total into a standard score using age-based normative data. The FSIQ-4 standard score ranges from 40 to 160. Higher scores represent better cognitive functioning and a score of <70 is used to determine intellectual disability.
  score on a scale | 74.71 (23.14) | 71.56 (24.40) | 73.16 (23.73)
Vineland Adaptive Behavior Scales (VABS-II) Expressive Communication [Mean (Standard Deviation); unit: score on a scale] — The VABS-II is a reliable and valid parent-report assessment of receptive, expressive, and written communication skills in individuals aged 3 to 22. Each item is scored as 0 (never), 1 (sometimes/partially), or 2 (usually), and these item scores are summed to produce a raw score, ranging from 0 to 108, then converted to a scale score using age-specific data. The Expressive Communication subdomain yields a v-scale score ranging from 1 to 24. Higher scale scores indicate better expressive communication skills and a raw score of 83 is equivalent to the expressive language of a four-year-old.
  score on a scale | 64.97 (29.15) | 63.63 (27.29) | 64.31 (28.15)
Sensory Over-Responsitivty (SensOR) Inventory Total [Mean (Standard Deviation); unit: units on a scale] — The SensOR Inventory is a 76-item caregiver-report measure of sensory processing patterns and sensitivities in individuals ages 3 or older. Items are scored with dichotomous yes/no responses. The scale consists of six domains (i.e., tactile, auditory, visual, olfactory, food texture, and movement-proprioceptive) that are summed for a total score. Scores range from 0-76 with higher scores indicate greater sensory over-responsiveness.
  units on a scale | 25.36 (12.95) | 29.46 (13.91) | 27.38 (13.54)
Child and Adolescent Symptom Inventory-4 Autism Anxiety Scale (CASI-Anx) [Mean (Standard Deviation); unit: score on a scale] — The CASI-Anx is a 20-item parent-report measure of anxiety in children with autism. Items are scored on a four-point Likert scale (i.e., 0-never, 1-sometimes, 2-often, 3-very often). The total score is calculated by taking the sum of the responses to all items. Scores range from 0 - 60 with higher scores indicating greater anxiety symptom severity.
  score on a scale | 18.55 (9.91) | 21.39 (10.47) | 19.95 (10.25)
Children's Fear Survey Schedule - Dental Subscale (CFSS-DS) [Mean (Standard Deviation); unit: score on a scale] — The CFSS-DS is a reliable and valid measure of dental fear in children. It is a 15-item, parent-report measure scored on a 5-point Likert scale (i.e., 1-not afraid at all to 5-very afraid). The total score is calculated by taking the sum of the responses to all items. Scores range from 15 -75 with higher scores indicating greater dental fear. Scores of 32-38 indicate borderline fear and those >38 suggest high dental fear.
  score on a scale | 45.94 (14.92) | 49.25 (12.10) | 47.57 (13.66)
Diagnoses [Count of Participants; unit: Participants] — Parent report of child diagnoses.
  Participants
    ADHD | 16 | 10 | 26
    Other Diagnoses | 27 | 27 | 54
Mother's education [Count of Participants; unit: Participants] — Parent report of mother's education.
  Participants
    <High school | 8 | 12 | 20
    High school | 12 | 10 | 22
    Some college of vocational | 28 | 27 | 55
    College degree | 22 | 19 | 41
Father's education [Count of Participants; unit: Participants] — Parent report of father's education.
  Participants
    <High school | 7 | 14 | 21
    High school | 21 | 15 | 36
    Some college or vocational | 18 | 13 | 31
    College degree | 17 | 16 | 33
    Not provided | 7 | 10 | 17

OUTCOME MEASURES:

1. Primary Outcome: Electrodermal Activity (EDA) - Skin Conductance Level (SCL)
Description: Electrodermal activity (EDA) is a non-invasive measure of the ability of the skin to conduct an electrical current, which increases when the sympathetic "fight or flight" nervous system is activated during times of stress.
Time Frame: Recorded continuously for three minutes prior to cleaning, through duration of cleaning (approximately 10-45 minutes), and for three minutes at end of cleaning for each dental cleaning.
Population: As this was a crossover study, all participants received cleanings in both the RDE and SADE conditions. Of the 162 participants, there were 248 analyzable observations for EDA SCLs.
Measure: Mean (Standard Deviation); unit: microsiemens (µS)
Groups:
- Sensory Adapted Dental Environment: In the Sensory Adapted Dental Environment the sensory characteristics of the dental environment are altered (visual, auditory, tactile adaptations).
  Sensory Adapted Dental Environment: The SADE intervention includes adaptations such as dimmed lighting, moving projections on the ceiling (fish, bubbles), exposure to soothing music, and application of a butterfly vest with wings that wrap around the child to provide calming sensations.
Arm/Group | Regular Dental Environment | Sensory Adapted Dental Environment
Number analyzed (Participants) | 127 | 121
microsiemens (µS) | 8.96 (5.29) | 7.74 (4.85)
Statistical Analysis 1: Comparison: Regular Dental Environment vs Sensory Adapted Dental Environment; Test type: Superiority; p = 0.01, Mixed-effects regression model; Adjusted for attained age and first or second clinic visit

2. Primary Outcome: Electrodermal Activity (EDA) - Non-specific Skin Conductance Responses (NS-SCR)
Description: Electrodermal activity (EDA) is a non-invasive measure of the ability of the skin to conduct an electrical current, which increases when the sympathetic "fight or flight" nervous system is activated during times of stress. Each unique increase >0.05uS in the EDA waveform is counted as an NS-SCR, indicating a increase in sympathetic nervous system activation; NS-SCRs are measured as a frequency per minute (calculated as the number of NS-SCRs/time).
Time Frame: as for outcome 1
Population: As this was a crossover study, all participants received cleanings in both the RDE and SADE conditions. Of the 162 participants, there were 245 analyzable observations for EDA NS-SCRs.
Measure: Mean (Standard Deviation); unit: number of NS-SCRs per minute (frequency)
Groups:
- Regular Dental Environment: There are two dental environments - the regular dental environment and the sensory dental environment; each child will be randomized to which is first. In the Regular dental environment, no sensory characteristics of the dental environment are altered, the cleaning is conducted as per usual.
- Sensory Adapted Dental Environment: In the Sensory Adapted Dental Environment, the sensory characteristics of the dental environment are altered (visual, auditory, tactile adaptations).
  Sensory Adapted Dental Environment: The SADE intervention includes adaptations such as dimmed lighting, moving projections on the ceiling (fish, bubbles), exposure to soothing music, and application of a butterfly vest with wings that wrap around the child to provide calming sensations.
Arm/Group | Regular Dental Environment | Sensory Adapted Dental Environment
Number analyzed (Participants) | 125 | 120
number of NS-SCRs per minute (frequency) | 4.25 (3.03) | 3.90 (2.72)
Statistical Analysis 1: Comparison: Regular Dental Environment vs Sensory Adapted Dental Environment; Test type: Superiority; p = 0.25, Mixed-effects regression model; Adjustment for attained age and first and second clinic visit

3. Secondary Outcome: Children's Dental Behavior Rating Scale (CDBRS)
Description: The CDBRS is a video-coded measure of overt distress behaviors exhibited by children during a routine dental visit. A research team member marks the presence or absence of three distress behaviors (mouth movement, head movement, forehead movement) and the presence or absence and the severity of two distress behaviors (whimper/cry/scream, verbal stall or delay) during each one-minute interval of a five-minute recording of a child receiving prophylaxis during their dental cleaning. Coding is conducted by a trained research team member who achieves strong inter-rater reliability with a second trained rater on a representative sample of children with and without ASD. Raw scores (range=0-45) are converted to a scale score ranging from 1 to 100, with higher scores indicating greater distress.
Time Frame: Videorecorded throughout dental cleaning (approximately 10-45 minutes); coded at a later time for the first five minutes of dental prophylaxis.
Population: As this was a crossover study, all participants received cleanings in both the RDE and SADE conditions. Of the 162 participants, there were 276 analyzable observations for CDBRS.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Regular Dental Environment | Sensory Adapted Dental Environment
Number analyzed (Participants) | 138 | 138
score on a scale | 46.41 (11.78) | 46.10 (10.77)
Statistical Analysis 1: Comparison: Regular Dental Environment vs Sensory Adapted Dental Environment; Test type: Superiority; p = 0.87, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Whimper, Cry, Scream Duration
Description: Duration of whimpers, cries, or screams, as scored by video coding.
Time Frame: Video-recorded throughout dental cleaning (approximately 10-45 minutes); coded at a later time for the first five minutes of dental prophylaxis.
Population: As this was a crossover study, all participants received cleanings in both the RDE and SADE conditions. Of the 162 participants, there were 276 analyzable observations for whimper, cry, scream duration.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Regular Dental Environment | Sensory Adapted Dental Environment
Number analyzed (Participants) | 138 | 138
minutes | 44.26 (68.39) | 19.70 (43.56)
Statistical Analysis 1: Comparison: Regular Dental Environment vs Sensory Adapted Dental Environment; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Whimper, Cry, Scream Frequency
Description: Frequency of whimpers, cries, or screams, as scored by video coding.
Time Frame: as for outcome 4
Population: As this was a crossover study, all participants received cleanings in both the RDE and SADE conditions. Of the 162 participants, there were 276 analyzable observations for whimper, cry, scream frequency.
Measure: Mean (Standard Deviation); unit: events
Arm/Group | Regular Dental Environment | Sensory Adapted Dental Environment
Number analyzed (Participants) | 138 | 138
events | 9.83 (9.96) | 6.02 (7.10)
Statistical Analysis 1: Comparison: Regular Dental Environment vs Sensory Adapted Dental Environment; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Mouth Movement Frequency
Description: Frequency of mouth movement impeding treatment, as scored by video coding.
Time Frame: as for outcome 4
Population: As this was a crossover study, all participants received cleanings in both the RDE and SADE conditions. Of the 162 participants, there were 276 analyzable observations for mouth movement frequency.
Measure: Mean (Standard Deviation); unit: events
Arm/Group | Regular Dental Environment | Sensory Adapted Dental Environment
Number analyzed (Participants) | 138 | 138
events | 5.43 (6.32) | 3.20 (4.15)
Statistical Analysis 1: Comparison: Regular Dental Environment vs Sensory Adapted Dental Environment; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Head Movement Frequency
Description: Frequency of head movement away from the dentist and/or equipment impeding treatment, as scored by video coding.
Time Frame: as for outcome 4
Population: As this was a crossover study, all participants received cleanings in both the RDE and SADE conditions. Of the 162 participants, there were 276 analyzable observations for head movement frequency.
Measure: Mean (Standard Deviation); unit: events
Arm/Group | Regular Dental Environment | Sensory Adapted Dental Environment
Number analyzed (Participants) | 138 | 138
events | 16.36 (19.39) | 11.68 (13.92)
Statistical Analysis 1: Comparison: Regular Dental Environment vs Sensory Adapted Dental Environment; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Faces Pain Scale - Revised
Description: The Faces Pain Scale - Revised is single-item self-report measure used to assess the perception and intensity of pain in children. The scale is comprised of six faces depicting increasing levels of pain ranging from a neutral expression (no pain) to a face showing severe pain. Each face corresponds to a numerical value on a 0-10 scale (0, 2, 4, 6, 8, 10). Higher scores indicate greater perception and intensity of pain.
Time Frame: Completed at the end of each dental cleaning (approximately 1-2 minutes)
Population: As this was a crossover study, all participants received cleanings in both the RDE and SADE conditions. Of the 162 participants, there were 114 usable scores for the Faces Pain Scale-Revised.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Regular Dental Environment | Sensory Adapted Dental Environment
Number analyzed (Participants) | 57 | 57
score on a scale | 2.37 (3.50) | 2.14 (3.13)
Statistical Analysis 1: Comparison: Regular Dental Environment vs Sensory Adapted Dental Environment; Test type: Superiority; p = 0.92, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Dental Sensory Sensitivity Scale
Description: The Dental Sensory Sensitivity Scale is a child-report measure assessing the presence and magnitude of discomfort with different sensory stimuli in the dental environment (i.e., tactile, auditory, proprioceptive). The scale is comprised of 6 items rated on a 3-point Likert scale ranging from 0 (not at all) to 2 (a lot). Scores range from 0 - 12 with higher scores indicating greater sensory discomfort during routine dental treatment.
Time Frame: Completed at the end of each dental cleaning (approximately 3 minutes)
Population: As this was a crossover study, all participants received cleanings in both the RDE and SADE conditions. Of the 162 participants, there were 106 usable scores for the Dental Sensory Sensitivity Scale.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Regular Dental Environment | Sensory Adapted Dental Environment
Number analyzed (Participants) | 53 | 53
score on a scale | 3.68 (3.06) | 3.06 (2.74)
Statistical Analysis 1: Comparison: Regular Dental Environment vs Sensory Adapted Dental Environment; Test type: Superiority; p = 0.16, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Anxiety and Cooperation Scale
Description: The Anxiety and Cooperation Scale (A & C Scale) has been shown to assess children's anxiety, fear, and cooperation as rated by dentists, and has good established reliability and validity. Following a routine dental cleaning, the dentist rated overall patient behavior during treatment using a one-item Likert scale ranging from 0 (relaxed, smiling, demonstrates desired behavior, complies with demands) to 5 (out of control, loud crying, reverts to primitive flight responses, physical restraint required).
Time Frame: Completed at the end of each dental cleaning (approximately 1 minute)
Population: As this was a crossover study, all participants received cleanings in both the RDE and SADE conditions. Of the 162 participants, there were 276 usable scores for the Anxiety and Cooperation Scale.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Regular Dental Environment | Sensory Adapted Dental Environment
Number analyzed (Participants) | 138 | 138
score on a scale | 2.03 (1.77) | 1.88 (1.61)
Statistical Analysis 1: Comparison: Regular Dental Environment vs Sensory Adapted Dental Environment; Test type: Superiority; p = 0.76, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Frankl Scale
Description: The Frankl Scale is dentist-report measure of a child's overall behavior during a dental visit. It is an observational, single-item measure that includes four behavioral categories, each assigned a numerical value (1=definitely negative, 2=negative, 3=positive, 4=definitely positive). Higher scores indicate greater cooperation and less distress.
Time Frame: Completed at the end of each dental cleaning (approximately 1 minute)
Population: As this was a crossover study, all participants received cleanings in both the RDE and SADE conditions. Of the 162 participants, there were 276 usable scores for Frankl Scale.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Regular Dental Environment | Sensory Adapted Dental Environment
Number analyzed (Participants) | 138 | 138
score on a scale | 2.61 (1.01) | 2.68 (0.98)
Statistical Analysis 1: Comparison: Regular Dental Environment vs Sensory Adapted Dental Environment; Test type: Superiority; p = 0.80, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: Duration
Description: The length of time to complete the dental cleaning. Used for cost-analysis of the intervention.
Time Frame: Time from beginning to end of dental cleaning (approximately 10-45 minutes); recorded for each visit
Population: As this was a crossover study, all participants received cleanings in both the RDE and SADE conditions. Of the 162 participants, there were 252 analyzable durations.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Regular Dental Environment | Sensory Adapted Dental Environment
Number analyzed (Participants) | 126 | 126
minutes | 10.51 (3.86) | 10.20 (4.14)
Statistical Analysis 1: Comparison: Regular Dental Environment vs Sensory Adapted Dental Environment; Test type: Superiority; p < 0.0001, Multivariate linear regression; Adjusted for autism severity, IQ, dental fear and anxiety, sensory over-responsivity, general anxiety, expressive communication, gender, and age

13. Secondary Outcome: Number of Hands Used to Restrain Child
Description: The maximum number of hands (at any one time) required to restrain the child during the dental cleaning experience was utilized as a measure of cost and also a measure of uncooperative behavior. This variable was recorded on researcher notes during the dental cleaning and was verified using the videotape of the dental cleaning. Scoring included presence/absence as well as the number of hands used for restraint purposes during the cleaning.
Time Frame: Recorded throughout the dental cleaning (approximately 10-45 minutes)
Population: As this was a crossover study, all participants received cleanings in both the RDE and SADE conditions. Of the 162 participants, there were 302 analyzable data points.
Measure: Mean (Standard Deviation); unit: hands
Arm/Group | Regular Dental Environment | Sensory Adapted Dental Environment
Number analyzed (Participants) | 153 | 149
hands | 2.14 (2.64) | 1.83 (2.32)
Statistical Analysis 1: Comparison: Regular Dental Environment vs Sensory Adapted Dental Environment; Test type: Superiority; p = 0.61, General linear mixed model

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for any reportable events throughout study completion. The duration of each participant's study participation was approximately 1 year.
Description: There were no occurrences of Serious Adverse Events, All-Cause Mortalities, or Other (Not Including Serious) Adverse Events throughout the duration of the study.
Arm/Group | Regular Dental Environment | Sensory Adapted Dental Environment
All-Cause Mortality (participants affected / at risk) | 0/151 | 0/150
Serious Adverse Events (participants affected / at risk) | 0/151 | 0/150
Other Adverse Events (participants affected / at risk) | 0/151 | 0/150

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-09-18): https://cdn.clinicaltrials.gov/large-docs/51/NCT02430051/Prot_SAP_000.pdf
  • Informed Consent Form (2019-11-19): https://cdn.clinicaltrials.gov/large-docs/51/NCT02430051/ICF_001.pdf